CLINICAL TRIAL: NCT00490698
Title: Bone-Targeted Therapy Combining Zoledronate With Atorvastatin in Renal Cell Carcinoma: A Phase II Study
Brief Title: Zoledronate With Atorvastatin in Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0652
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Cancer; Renal Cell Carcinoma
Keywords: Kidney Cancer; Renal Cell Carcinoma; Bone-Targeted Therapy; Zoledronate; Zometa; Atorvastatin; Lipitor; RCC
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Zoledronic Acid; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zoledronate + Atorvastatin (Experimental): Zoledronate 4 mg intravenous (IV) once every 4 Weeks + Atorvastatin 20 mg orally (PO) daily
  Interventions: Drug: Zoledronate; Drug: Atorvastatin

INTERVENTIONS:
Drug: Zoledronate — 4 mg IV Once Every 4 Weeks
  Other Names: Zometa
Drug: Atorvastatin — 20 mg PO Daily
  Other Names: Lipitor

SUMMARY:
Objectives:

Primary:

Evaluate clinical outcome based on the time to skeletal events after bone-targeted therapy

Secondary:

1. Evaluate clinical outcome based on the presence of calcification at the site of osteolytic metastases
2. Measure bone-formation and resorption markers at baseline and during bone-targeted therapy.
3. Assess effect of the bone-targeted regimen on serum cholesterol levels

DETAILED DESCRIPTION:
Kidney cancer often spreads (metastases) to the bones. Zoledronate is designed to protect the bones from pain and from breaking as a result of cancer. Atorvastatin is a drug that lowers cholesterol levels in the blood. Combining these medications may make zoledronate more effective.

If you are found to be eligible to take part in this study, you will be given zoledronate intravenously (IV--through a needle in your vein) over fifteen minutes,1 time every 4 weeks. You will take a pill, atorvastatin, by mouth once time a day every day that you are on the study. Every 4 weeks is considered 1 study "cycle".

You will need to return to M. D. Anderson for check-ups every 8 -12 weeks. Urine will be collected for routine tests. You will have x-rays, bone scans, and/or CT scans to check on the status of the disease.

You will receive at least 2 cycles of treatment unless intolerable side effects occur or your disease gets worse. You may receive more than 2 cycles if you are benefitting from the study drugs.

You will be followed every 8 weeks for up to 1 year for skeletal events (symptoms related to disease moving to or getting worse in your bones). You will be taken off study if you experience a skeletal event or at the end of the 1-year monitoring period. Monitoring may be done with a local doctor or at M. D. Anderson. No extra testing or procedures are needed during this period.

This is an investigational study. The combination of the 2 drugs given in this study is investigational for the treatment of bone metastases. Zoledronate is approved for the treatment of bone metastases. Atorvastatin has been approved by the FDA for lowering cholesterol. About 38 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed renal cell carcinoma
2. Must have evidence of predominant bone metastases on X-rays, bone scan, MRI or CT scan. No requirement for bidimensionally measurable lesions.
3. Impending complications (such as pathological fractures and spinal cord compressions) from skeletal metastases must be controlled by surgery or radiation therapy.
4. Patients with prior or on concurrent immunotherapy or chemotherapy are eligible, excluding those on drugs that will interact with statins (Cytochrome P450 2C9 Pathway).
5. Patients with prior or concurrent treatment with bisphosphonates or statins are eligible.
6. Patients with hypercalcemia are eligible.
7. Adequate physiologic reserves as evidenced by:Zubrod performance status of </= 2; Transaminase and conjugated bilirubin less than twice the upper limit of normal; Creatinine Clearance >/= 30 ml/min.
8. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study.

Exclusion Criteria:

1. Patients of childbearing potential not practicing adequate contraception.
2. Patients with poor dentition or recent major dental procedures.
3. History of other malignancies other than non-melanoma skin cancer or carcinoma-in-situ of the cervix unless in complete remission and off therapy for that disease for at least 5 years.
4. Overt psychosis or mental disability or otherwise incompetent to give informed consent.
5. Known hypersensitivity to Zometa (zoledronic acid), other bisphosphonates, or to fluvastatin.
6. Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
7. Recent (within 6 weeks) or planned dental or jaw surgery (e.g., extraction, implants)
8. Active liver disease or unexplained persistent elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times upper limits of normal (ULN)
9. Serum creatine kinase (CK) > 3 times ULN
10. Patients taking concurrent agents that may increase risk of myopathy such as fibric acid derivatives, nicotinic acid, cyclosporine, azole antifungals (itraconazole, ketoconazole, and fluconazole), macrolide antibiotics (erythromycin, clarithromycin, HIV protease inhibitors, nefazodone, delavirdine, cyclosporine, and grapefruit juice.
11. History of alcohol abuse as such condition independently predisposes patients to myopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ming Tu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Manoukian GE, Tannir NM, Jonasch E, Qiao W, Haygood TM, Tu SM. Pilot trial of bone-targeted therapy combining zoledronate with fluvastatin or atorvastatin for patients with metastatic renal cell carcinoma. Clin Genitourin Cancer. 2011 Dec;9(2):81-8. doi: 10.1016/j.clgc.2011.07.001. Epub 2011 Oct 1. PMID 21958521
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 1, 2006 to January 31, 2008. All recruitment done at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Zoledronate + Atorvastatin
Started | 11
Completed | 1
Not Completed | 10
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 7
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Zoledronate + Atorvastatin
Number analyzed (Participants) | 11
Age Continuous [Median (Full Range); unit: years] | 56.6 [42 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Median Time to First Skeletal-related Event
Description: Time to skeletal events, defined as a metastatic site requiring radiotherapy or any surgical intervention (eg, embolization, radiofrequency ablation, intrathecal catheter placement) or complications from skeletal metastatic lesions (eg, pathologic fracture, spinal cord compression). Time to skeletal events monitored every 8 weeks for at least 1 year.
Time Frame: Up to 1 year
Population: Four participants did not experience skeletal events.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zoledronate + Atorvastatin
Number analyzed (Participants) | 7
months | 9 [4.1 to 18.1]

ADVERSE EVENTS:
Time Frame: 4 years and 3 months
Description: "Definitely" and "Probably" related World Health Organization (WHO)classification grade 1 and 2 adverse events were reported.
Arm/Group | Zoledronate + Atorvastatin
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronate + Atorvastatin (N=11)
Transient ischemic attack (Blood and lymphatic system disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronate + Atorvastatin (N=11)
Desquamatory rash (Skin and subcutaneous tissue disorders) | 1
Fever (Infections and infestations) | 1
Fatigue (General disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No